CLINICAL TRIAL: NCT05913921
Title: A Randomized, Open-label, Single-dose, Two-preparation, Two-period, Two-sequence Bioequivalence Study Between Amphotericin B Liposome for Injection and AmBisome® in Healthy Subjects
Brief Title: Bioequivalence of Amphotericin B Liposome for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HC1507-004
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Amphotericin B; Injections; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Experimental): 16 healthy subjects assigned to the sequence TR were administrated intravenously for 120 mins with the test product of amphotericin B liposome for injection in period 1 and the reference product of AmBisome® in period 2
  Interventions: Drug: Amphotericin B liposome for injection; Drug: AmBisome
- Sequence RT (Experimental): 16 healthy subjects assigned to the sequence RT were administrated intravenously for 120 mins with the reference product of AmBisome® in period 1 and the test product of amphotericin B liposome for injection in period 2
  Interventions: Drug: Amphotericin B liposome for injection; Drug: AmBisome

INTERVENTIONS:
Drug: Amphotericin B liposome for injection — IV infusion, 2.0 mg/kg
  Other Names: the test product
Drug: AmBisome — IV infusion, 2.0 mg/kg
  Other Names: the reference product

SUMMARY:
The main purpose of this study is to evaluate the bioequivalence of two different amphotericin B liposome for injection after single IV infusion at the same dose in normal healthy subjects.

DETAILED DESCRIPTION:
Single-Center, Open-Label, Randomized, Two-treatment, Crossover, Two-sequence, Single-Dose Bioequivalence study of Amphotericin B Liposome for Injection and AmBisome (Amphotericin B) Liposome for Injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give informed consent before the trial, fully understand the content, process and possible adverse reactions, and voluntarily sign a written informed consent.
2. The subjects can communicate well with the investigators and complete the trial according to protocol.
3. Sex: male or female subjects.
4. Age of 18 - 55 years (inclusive).
5. BMI: 18.6-28.5 kg/m^2 (inclusive), with a minimum weight of 50 kg (inclusive) for males and 45 kg (inclusive) for females.

Exclusion Criteria:

1. Allergic constitution, or known history of allergy to the components of the study drug or similar drugs.
2. Subjects with the following diseases of clinical significance (including but not limited to diseased related to respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin system, psychiatric system, otorhinolaryngology).
3. Subjects with liver and kidney diseases that affect the pharmacokinetic of drugs.
4. Those who underwent major surgery within 6 months prior to initial administration, or who planned to undergo surgery during the study.
5. Clinically significant abnormalities in vital signs, physical examination, electrocardiogram and laboratory examination (including but not limited to alanine aminotransferase (ALT) or aspartate aminotransferase (AST) and creatinine above the upper limit of normal).
6. Subjects with a history of hepatitis B, hepatitis C, AIDS, syphilis and/or abnormalities in one or more of the four tests for infectious diseases with clinical significance.
7. Blood loss or blood donation of more than 200 mL within 3 months prior to initial administration (except for female menstrual period), and/or platelet donation within 2 weeks prior to initial administration.
8. Use of any drug within 14 days prior to initial administration (except for topical drugs with local effects).
9. Use of any investigational medicinal product within 3 months prior to initial administration.
10. A history of drug abuse, and/or drug use within 3 months prior to screening, and/or habitual use of any drug, including Chinese herbs.
11. Positive urine drug screening.
12. Those who smoked more than 5 cigarettes per day within 3 months prior to screening and/or did not agree to refrain from using any tobacco products during hospitalization.
13. Regular drinkers within 6 months prior to screening, i.e., those who drank more than 14 units of alcohol per week, and/or those who could not stop drinking alcohol during their hospitalization, and/or test positive for breath alcohol.
14. Those who consume excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day, and/or do not agree that tea, coffee and/or caffeinated foods, grapefruit (grapefruit) and/or grapefruit juice (grapefruit juice), and/or products containing opium poppy are prohibited during hospitalization.
15. Those who have a birth plan (including sperm donation and egg donation) and/or do not agree to take effective contraceptive methods (non-drug during the trial period) within 3 months after signing informed consent form.
16. Subjects who may not be able to complete the study for other reasons or who the investigator considers should not be included.

    In addition to the above requirements, female subjects who meet the following conditions shall also be excluded:
17. Pregnant or lactating women or those with positive pregnancy results.
18. Those who have used oral contraceptives within 30 days prior to initial administration.
19. Use of long-acting estrogen and/or progesterone injections and/or implants within 6 months prior to initial administration.
20. Women of childbearing age who have unprotected sex with their partner within 14 days prior to initial administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | predose to 216 hours post dose
  90% CI of Cmax of liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%
Bioequivalence based on AUC0-t | predose to 216 hours post dose
  90% CI of AUC0-t of liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%
Bioequivalence based on AUCinf | predose to 216 hours post dose
  90% CI of AUC0-∞ of liposome-encapsulated and non-liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%

SECONDARY OUTCOMES:
Cmax | predose to 216 hours post dose
  90% CI of Cmax of non-liposome-encapsulated and total Amphotericin B
AUC0-t | predose to 216 hours post dose
  90% CI of AUC0-t of non-liposome-encapsulated and total Amphotericin B
AUC0-∞ | predose to 216 hours post dose
  90% CI of AUC0-∞ of non-liposome-encapsulated and total Amphotericin B

CONTACTS AND LOCATIONS:
Overall Officials: XiaoAi He, Principal Investigator — Haikou People's Hospital
Locations (1):
- Haikou people's Hospital, Haikou, Hainan, China